CLINICAL TRIAL: NCT06888076
Title: An Observational Study to Assess the Safety of Pertagen®, a Recombinant Acellular Pertussis Vaccine in Pregnant Women in Thailand
Brief Title: Study Evaluating the Safety of a Recombinant Acellular Pertussis Vaccine in Pregnant Women
Status: Active, not recruiting | Type: Observational
Sponsor: BioNet-Asia Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PerMIS-01
Record Dates: First submitted 2025-03-12; First posted 2025-03-21 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Pertussis Vaccines; Pertussis (Whooping Cough)
Keywords: Pertussis; whooping cough
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women received Pertagen® and have given birth in Jan 2021-Apr 2024 and their infants: The pregnant women (previously vaccinated with Pertagen®) and have given birth in Thailand from Jan 2021 - Apr 2024 and infants born to pregnant women who received Pertagen®.

SUMMARY:
This is an observational, retrospective, cohort, safety study in pregnant women (vaccinated with Pertagen®) and have given birth in Thailand from January 2021 to April 2024 and infants born to pregnant women who received Pertagen®.

Following approval of the final protocol from the Institutional Review Board (IRB) and/or Ethics Committee (EC) and written approval from hospital directors/medical doctors as per requirements of each institutions. The assigned Ob-gyn specialist/physician at each study site will review the medical record of pregnant women (January 2020 to April 2024) based on study selection criteria. Safety information of pregnant women who received Pertagen® and have given birth from January 2021 to April 2024 and infants born to pregnant women who received Pertagen® will be obtained from medical records in hospitals/clinics and will be reported in case report form (CRF) by assigned Ob-gyn specialist/physician at each study site. The assigned Ob-gyn specialist/physician at each study site who will review the medical records and report the data in case report form (CRF) is not part of the research team.

DETAILED DESCRIPTION:
A CRF has been developed and will be used to collect safety information on pregnancy outcomes including the health status of infants at birth. The following definitions will be used for data collection

* The 2nd trimester of pregnancy is defined as gestational period between 13-26 weeks
* The 3rd trimester of pregnancy is defined as gestational period from 27 weeks to delivery.
* Full term birth is defined as delivery of a baby at gestational age (GA) ≥37 weeks.
* Preterm birth is defined as delivery of a baby at GA<37 weeks.
* Complications during delivery may include postpartum hemorrhage, maternal fever or infection, or any maternal and fetal indications that may require emergency caesarean section.
* Safety information of pregnancy and delivery outcome refers to health of women during pregnancy and childbirth (WHO 2024). The most common direct causes of maternal injury and death are excessive blood loss, infection, high blood pressure, unsafe abortion, and obstructed labor, as well as indirect causes such as anemia and heart disease (WHO 2024).
* A newborn is defined as healthy at birth if discharged from the hospital in the first few days of life.
* A newborn is defined as not healthy if with difficulty of breathing, congenital abnormality or other conditions that would require prolonged stay at the hospital.

To ensure the privacy and confidentiality of the collected data, strict adherence to all relevant data protection regulations will be followed.

ELIGIBILITY:
Inclusion Criteria:

1. Data of pregnant women previously vaccinated with Pertagen® during second or third trimester of pregnancy and have given birth in Thailand from January 2021 to April 2024 and infants born to pregnant women who received Pertagen® during pregnancy.
2. Infant of pregnant women who received Pertagen® during second or third trimester of pregnancy

Exclusion Criteria:

1. pregnant women previously vaccinated with Pertagen®, but maternal and infant data at delivery/birth cannot be obtained.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The pregnant women who received Pertagen® and have given birth from January 2021 to April 2024 and infants born to pregnant women who received Pertagen® which obtained from medical records in hospitals/clinics
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
1 Number and percentage of pregnant women vaccinated with Pertagen who had experienced full term and preterm (or premature) delivery 1.2 Number and percentage of pregnant women vaccinated with Pertagen® who had experienced complications during delivery. | Safety profile of Pertagen® in pregnant women at delivery
  * Full term birth is defined as delivery of a baby at gestational age (GA) ≥37 weeks.
  * Preterm birth is defined as delivery of a baby at GA<37 weeks.
  * Complications during delivery may include postpartum hemorrhage, maternal fever or infection, or any maternal and fetal indications that may require emergency caesarean section.

SECONDARY OUTCOMES:
1 Number and percentage of healthy infants born to mothers who received Pertagen® during pregnancy. 2.2 Number and percentage of not healthy infants born to mothers who received Pertagen® during pregnancy | Safety profile of Pertagen® in infants born to mother who received Pertagen® at birth
  * A newborn is defined as healthy at birth if discharged from the hospital in the first few days of life.
  * A newborn is defined as not healthy if with difficulty of breathing, congenital abnormality or other conditions that would require prolonged stay at the hospital.

OTHER OUTCOMES:
Number and percentage of pregnant women had experienced preterm (or premature) delivery in pregnant women received Pertagen® and gave birth during January 2021 - April 2024 and in pregnant women received licensed Td vaccine and gave during 2019-2020 | 1. Data from review medical records of pregnant women who received Pertagen® and have given birth in Jan 2021 - Apr2024 with their infants. 2. - Data of pregnant women received Td vaccine and gave birth in 2019-2020 (source: HDC, MopH Thailand)
  Preterm birth is defined as delivery of a baby at GA<37 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Soaud Mansouri, PhD., Study Director — Bionet-Asia Co., Ltd (Branch1)
Locations (1):
- Faculty of Medicine Siriraj Hospital Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No